CLINICAL TRIAL: NCT02958969
Title: Apixaban for Primary Prevention of Venous Thromboembolism in Patients With Multiple Myeloma Receiving Immunomodulatory Therapy
Brief Title: Apixaban for Primary Prevention of Venous Thromboembolism in Patients With Multiple Myeloma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gregory Piazza (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Gregory Piazza, Sponsor Investigator, Brigham and Women's Hospital
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 18-493
Record Dates: First submitted 2016-11-05; First posted 2016-11-08 (Estimated); Results first posted 2019-12-06 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Venous Thromboembolism; Multiple Myeloma
Keywords: venous thromboembolism; multiple myeloma; anticoagulation
MeSH Terms: conditions — Venous Thromboembolism; Multiple Myeloma | interventions — apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Apixaban (Experimental): apixaban 2.5 mg orally twice daily for primary prevention of VTE for a duration of 6 months
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban — apixaban 2.5 mg orally twice daily for primary prevention of VTE for a duration of 6 months
  Other Names: Thromboprophylaxis

SUMMARY:
Patients living with multiple myeloma (MM) have an increased risk of venous thromboembolism (VTE) due to the disease itself and the use of targeted therapies, including immunomodulatory drugs (IMiDs). Prevention of VTE has become a major management challenge during MM treatment. There is a paucity of data with respect to the non-vitamin K oral anticoagulants (NOACs) in the cancer population. However, the NOACs offer comparable efficacy but improved safety compared with warfarin. Apixaban has shown excellent safety and efficacy for treatment and prevention of recurrent VTE (1,2). The safety and efficacy of apixaban for primary prevention of VTE in MM patients has not been established.

Aim #1: To quantify the 6-month rate of major and clinically relevant non-major bleeding in MM patients receiving IMiDs who are prescribed apixaban 2.5 mg orally twice daily for primary prevention of VTE.

Hypothesis #1: The 6-month rate of major and clinically relevant non-major bleeding in MM patients receiving IMiDs who are prescribed apixaban 2.5 mg orally twice daily for primary prevention of VTE will be ≤3% (2). Although the MM population, in general, has a higher medical acuity than that of the previous large randomized controlled trials of apixaban, we will be selecting a stable population of MM patients who are appropriate for immunomodulatory therapy.

Aim #2: To quantify 6-month rate of symptomatic VTE in MM patients receiving IMiDs who are prescribed apixaban 2.5 mg orally twice daily for primary prevention of VTE.

Hypothesis #2: The 6-month rate of symptomatic VTE in MM patients receiving IMiDs who are prescribed apixaban 2.5 mg orally twice daily for primary prevention of VTE will be <7% (3). Although additional therapies for MM such as dexamethasone and erythropoietin-stimulating agents may further increase the risk of VTE, the rate of incident VTE should be reduced to <7% with apixaban.

DETAILED DESCRIPTION:
MM is associated with an increased risk of venous thromboembolism (VTE). The use of targeted therapies, including immunomodulatory drugs (IMiDs), has improved outcomes for patients with MM but also increases the risk of VTE. Prevention of VTE has become a major management dilemma during MM treatment. There is a paucity of data with respect to the non-vitamin K oral anticoagulants (NOACs) in the cancer population, including patients with MM. However, the NOACs have been shown to offer comparable efficacy but improved safety compared with warfarin. Apixaban has shown excellent safety and efficacy for treatment and prevention of recurrent VTE (1,2). Compared with injectable thromboprophylactic regimens such as enoxaparin, apixaban offers the advantages of being orally administered and less reliant on renal clearance. The safety and efficacy of apixaban for primary prevention of VTE in MM patients has not been established. The current study will evaluate apixaban (2.5 mg twice daily) in a patient population without a history of prior VTE. Although the current study population is high risk for VTE, it is likely to be lower risk for VTE than those of the prior randomized controlled trials of apixaban for secondary prevention. Furthermore, current practice is to provide MM patients receiving IMiDs with prophylactic doses (not treatment doses) of low-molecular weight heparin (such as enoxaparin 40 mg injected daily). Accordingly, the rationale to test apixaban (2.5 mg twice daily) is consistent with the standard practice of prophylactic anticoagulation.

The current study will provide event rates that will inform the design of a larger randomized controlled trial. If safe and effective, apixaban will satisfy a critical unmet need and will represent a substantial advance and "game changer" in the prevention of VTE in this high risk patient population.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Age > 18 years
* Current or prior diagnosis of symptomatic MM based on International Myeloma Working Group (IMWG) guidelines (http://imwg.myeloma.org/category/guidelines-2/) and will be starting or already receiving IMiD therapy with thalidomide [Thalomid], lenalinomide [Revlimid], or pomalidomide [Pomalyst]
* IMiD therapy given in the setting of newly diagnosed MM, relapsed MM, progressive MM, maintenance therapy or consolidation therapy as per IMWG criteria
* Willing to provide written informed consent
* Eastern Cooperative Oncology Group (ECOG) functional status ≤ 2
* Providers must plan to treat the patient with IMiD therapy for a minimum of 6 cycles

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Women of child-bearing potential who are unwilling or unable to use an acceptable method of birth control (such as oral contraceptives, other hormonal contraceptives [vaginal products, skin patches, or implanted or injectable products], or mechanical products such as an intrauterine device or barrier methods [diaphragm, condoms, spermicides]) to avoid pregnancy for the entire study
* Any prior venous thromboembolism
* Contraindication to anticoagulant therapy
* Conditions for which serious bleeding may occur including:

  1. Current or within last 6 months: intracranial bleeding, intraocular bleeding, gastrointestinal bleeding, endoscopically documented ulcer disease
  2. Current or within last month: head trauma or other major trauma, major surgery
  3. Current or within last 2 weeks: stroke, neurosurgical procedure
  4. Current: gross hematuria, major unhealed wound, major surgery planned during the trial period, intracranial mass, vascular malformation, or aneurysm, overt bleeding, blood dyscrasia
  5. CNS involvement of MM or other history of CNS malignancy
* Active and clinically significant liver disease
* Uncontrolled hypertension: systolic blood pressure >180 mm Hg or diastolic blood pressure >100 mm Hg
* Current endocarditis
* Requirement for ongoing anticoagulant therapy, including mechanical heart valve replacement and atrial fibrillation
* Severe valvular heart disease, including rheumatic heart disease and mitral stenosis
* Bioprosthetic heart valve replacement
* Requirement for dual antiplatelet therapy or single agent antiplatelet therapy with clopidogrel, prasugrel, or ticagrelor
* Requirement for aspirin at a dose higher than 165 mg daily.
* Hemoglobin < 9 mg/dL at time of screening
* Platelet count < 100,000/mm3 at time of screening
* Serum calculated creatinine clearance (CrCl) < 25 ml/m at time of screening
* Alanine aminotransferase or aspartate aminotransferase level > 2 times the upper limit of the normal at time of screening
* Total bilirubin level > 1.5 times the upper limit of the normal at time of screening
* Life expectancy < 12 months or hospice care
* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness
* Receiving concurrent non-FDA-approved or investigational agents or has received an investigational agent within the past 30 days prior to the first dose of study treatment (with the exception of approved medications being used for an approved indication, e.g., investigating a new dosing regimen for an approved indication).
* Any condition, which in the opinion of the investigator, would put the subject at an unacceptable risk from participating in the study
* Any other medical, social, logistical, or psychological reason, which in the opinion of the investigator, would preclude compliance with, or successful completion of, the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-11-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Vanderbilt University Medical Center, Nashville, Tennessee

REFERENCES:
- [Derived] Kahale LA, Matar CF, Tsolakian I, Hakoum MB, Yosuico VE, Terrenato I, Sperati F, Barba M, Hicks LK, Schunemann H, Akl EA. Antithrombotic therapy for ambulatory patients with multiple myeloma receiving immunomodulatory agents. Cochrane Database Syst Rev. 2021 Sep 28;9(9):CD014739. doi: 10.1002/14651858.CD014739. PMID 34582035

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Apixaban
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Apixaban
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 42
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [51 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 41
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Symptomatic Venous Thromboembolism
Description: Symptomatic deep vein thrombosis or pulmonary embolism
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban
Number analyzed (Participants) | 50
Participants | 0

2. Primary Outcome: Frequency of Major and Clinically Relevant Non-major Bleeding
Description: Major and clinically relevant non-major bleeding. Using the ISTH classification, bleeding is defined as major if it is overt and associated with a decrease in the hemoglobin level of 2 g/dL or more, requires the transfusion of 2 or more units of blood, occurs into a critical site, or contributes to death (12).
  Using the ISTH classification, clinically relevant nonmajor bleeding is defined as overt bleeding not meeting the criteria for major bleeding but associated with medical intervention, surgical intervention, or interruption of the study drug.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban
Number analyzed (Participants) | 50
Participants | 3

3. Secondary Outcome: Frequency of All-cause Mortality
Description: All-cause mortality at 6 months will be recorded. Cause of death will be classified as related to cancer, myocardial infarction, PE, other cardiovascular or other disease state. Death will be attributed to PE if there is evidence to support an association with PE.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban
Number analyzed (Participants) | 50
Participants | 0

4. Secondary Outcome: Frequency of Atherothrombotic Events
Description: 6-month rates of myocardial infarction and stroke will be calculated.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban
Number analyzed (Participants) | 50
Participants | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Apixaban
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 3/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apixaban (N=50)
non-major bleeding (Blood and lymphatic system disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
The study is limited by small sample size. The study included 10 patients receiving IMiD monotherapy for maintenance which are patients at lowest risk for VTE due to the absence of dexamethasone and low disease burden.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-08): https://cdn.clinicaltrials.gov/large-docs/69/NCT02958969/Prot_SAP_000.pdf